CLINICAL TRIAL: NCT04815655
Title: Cartilage Tympanoplasty for Recurrent Perforation Full Thickness Versus Partial Thickness Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Caroleen Mounir Tawfik, principle investigator, Assiut University
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cartilage tympanoplasty
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Cartilage Tympanoplasty

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cartilage tympanoplasty — is the reconstruction of the tympanic membrane (TM) by using catilage

SUMMARY:
Cartilage tympanoplasty for recurrent perforation full thickness versus partial thickness graft.

DETAILED DESCRIPTION:
To compare between outcomes of full thickness versus partial thickness graft in cartilage tympanoplasty using cartilage slicer

ELIGIBILITY:
Inclusion Criteria:

1 -patients with safe chronic suppurative otitis media 2- patients with recurrent perforations 3- patients with conductive hearing loss- 4- patients above 18 years

Exclusion Criteria:

1. active infection
2. sensorineural hearing loss
3. compromised immune system 4 - patients age below 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
To compare between outcomes of full thickness versus partial thickness graft in cartilage tympanoplasty using cartilage slicer | 1 year
  To compare between outcomes of full thickness versus partial thickness graft in cartilage tympanoplasty using cartilage slicer

CONTACTS AND LOCATIONS:
Overall Officials: Hamza Elshafie, Professor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No